CLINICAL TRIAL: NCT06730711
Title: Association Between Blood Pressure and the Risk of Post-stroke Cognitive Impairment: a Retrospective Cohort Study
Brief Title: Association Between Blood Pressure and Risk of PSCI
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dingqun Bai, Director of rehabilitation Medicine, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 20241202
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Cognitive Decline; Blood Pressure
Keywords: stroke; cognitive impairment; blood pressure
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NPSCI: NPSCI was defined as a score of MMSE≥26.
- PSCI: The prime outcome PSCI was defined as the cognitive impairment occurred after stroke and was still present three months after stroke and cognitive impairment was defined as a score of MMSE<26.

SUMMARY:
This retrospective cohort study was designed to explore the relationship between blood pressure and cognitive impairment after stroke

DETAILED DESCRIPTION:
Patients who have been followed up for more than 3 months after stroke will be included in the study. Basic data of patients and factors that may be related to cognitive impairment will be collected, and the relationship between blood pressure and cognitive impairment after stroke will be explored by univariate regression analysis and multivariate regression analysis. Univariate logistic regression model and multivariate logistic regression model were used to explore the relationship between blood pressure level and the risk of cognitive impairment after stroke, and the effect of blood pressure level and cognitive impairment sub-line in different patients was evaluated by subgroup analysis.

ELIGIBILITY:
Inclusion criteria:

1. Patient diagnosed with stroke by CT or MRI,
2. Patients completed the MMSE scale at least once during hospitalization
3. The follow-up time was more than three months after the stroke occurred;

Exclusion criteria:

1. Patients with incomplete data, follow-up time less than three months after the stroke occurred less than 3 months,
2. Patients with pre-existing cognitive impairment before stroke according to their medical records,
3. patients failed to complete MMSE assessment because of aphasia or any other reasons,
4. Patients combined with malignant tumors, patients combined with psychiatric disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients admitted to the First Branch of the First Affiliated Hospital of Chongqing Medical University between 2022 and 2024 were retrospectively reviewed.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mental State Examination Scale (MMSE) | Mini-Mental State Examination (MMSE) assessment will be completeed at 3 monthes after stroke
  Global cognitive function assessment. Easy to use and one of the most used scales to screen person with cognitive impairment in the world. The minimum and maximum values range from 0 to 30. Higher score means better cognition level.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided